CLINICAL TRIAL: NCT06204094
Title: Total Neoadjuvant CAPOX and PD-1 Inhibitor（Sintilimab） Combined with Node-sparing Short-course Radiotherapy for MSS Locally Advanced of Middle and Low Rectal Cancer(CASINOs): an Open Label, Single-arm, Prospective Clinical Trial
Brief Title: Node-sparing Radiotherapy Combined with Total Neoadjuvant CAPOX and Sintilimab for MSS Middle and Low Rectal Cancer
Acronym: CASINOs
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Jinhua Central Hospital (Other)
Responsible Party: Principal Investigator, Cheng Cai, Clinical Professor, Jinhua Central Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Jinhua CH
Record Dates: First submitted 2024-01-02; First posted 2024-01-12 (Actual); Last update posted 2025-01-07 (Actual); Status verified 2025-01

CONDITIONS: Locally Advanced Rectal Cancer
Keywords: rectal cancer; microsatellite stability; node-sparing; CAPOX; radiotherapy; sintilimab; immunotherapy; neoadjuvant
MeSH Terms: conditions — Rectal Neoplasms | interventions — sintilimab; Capecitabine; Oxaliplatin

STUDY DESIGN:
Intervention Model Description: Radiation: node-sparing short-course radiotherapy (5Gy*5d) Drug: PD-1 antibody (Sintilimab) Drug: Capecitabine Drug: Oxaliplatin
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment Arm (Experimental): Participants will receive 5*5Gy node-sparing short-course radiation (radiation targeting the tumor bed without irradiating surrounding tumor-draining lymph nodes) concurrently with total neoadjuvant CAPOX and sintilimab regimens: Oxaliplatin, 130mg/m2, intravenous infusion,d1 of each cycle; Capecitabine, 1000mg/m2, PO, BID, d1-14 and sintilimab, 200mg intravenous infusion d1 of each cycle. CAPOX and sintilimab are repeated every 3 weeks for 8 cycles. Patients with cCR will be managed with a WW strategy, and patients who did not achieve cCR will receive TME surgery.
  Interventions:
  * Radiation: node-sparing short-course radiation
  * Drug: PD-1 antibody (Sintilimab)
  * Drug: Capecitabine
  * Drug: Oxaliplatin
  Interventions: Radiation: node-sparing short-course radiotherapy; Drug: Sintilimab; Drug: Capecitabine; Drug: Oxaliplatin; Procedure: TME surgery; Procedure: watch and wait

INTERVENTIONS:
Radiation: node-sparing short-course radiotherapy — 5Gy*5d, radiation targeting the tumor bed without irradiating surrounding tumor-draining lymph nodes
Drug: Sintilimab — 200mg intravenous infusion d1 of each cycle*8cycles
  Other Names: IBI308
Drug: Capecitabine — 1000mg/m2, PO, BID, d1-14 of each cycle*8cycles
Drug: Oxaliplatin — 130mg/m2, intravenous infusion,d1 of each cycle*8cycles
Procedure: TME surgery — laparoscopic or robotic TME surgery for non-cCR patients
  Other Names: total mesorectal excision
Procedure: watch and wait — WW for cCR patients
  Other Names: WW

SUMMARY:
phase II clinical trial to evaluate node-sparing short-course radiation combined with total neoadjuvant CAPOX and Sintilimab for MSS locally advanced rectal cancers.

DETAILED DESCRIPTION:
This is an open-label, prospective, single-center phase II clinical trial to evaluate node-sparing short-course radiation (Radiation targeting the tumor bed without irradiating surrounding tumor-draining lymph nodes) combined with total neoadjuvant CAPOX and PD-1 Inhibitor (Sintilimab) for patients with MSS locally advanced of middle and low rectal cancer. A total of 47 patients will be enrolled in this trial. The primary endpoint is the complete response(CR) rate, which includes cCR and pCR. The organ preservation rate, tumor regression grade, 3-year DFS, 3-year OS, and adverse effects will also be analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have a strong willingness to preserve the anus and are willing to receive neoadjuvant therapy.
* Male or Female aged 18-75.
* Patients diagnosed with low rectal cancer within 10 cm from the lower edge of the tumor to the anal verge by pelvic MRI and anorectoscopy, the clinical stage is cT2N+M0/cT3-4aN0/+M0, the lymph nodes are limited to the mesorectum, the circumferential resection margin is negative.
* Histologically confirmed rectal adenocarcinoma; Genetic testing suggests MSI-L or MSS, or tumor biopsy immunohistochemistry reveals pMMR, that is, MSH1, MSH2, MSH6, and PMS2 are all positive.
* Eastern Cooperative Oncology Group (ECOG) 0-1.
* No previous treatment(including anti-tumor therapy、immunotherapy or pelvic radiation).
* Adequate hematologic, hepatic, renal, thyroid and cardiac function: white blood cells ≥3500/mm3, neutrophils ≥1800/mm3, platelets ≥100,000/mm3, hemoglobin ≥100 g/L; activated partial thromboplastin time, prothrombin time and international normalized ratio ≤1.5 × ULN; aspartate aminotransferase and alanine aminotransferase ≤3.0 × upper limit of normal (ULN), bilirubin ≤1.25 × ULN, serum albumin ≥28 g/L. creatinine clearance ≥50 mL/mi, creatinine ≤1.5 × ULN;
* Informed consent form signed.

Exclusion Criteria:

* Patients with a previous history of malignant tumors besides rectal cancer.
* Patients with distant metastases before enrollment.
* Patients with positive internal or external iliac lymph nodes are assessed by MRI or CT.
* Patients with obstruction, perforation, or bleeding that require emergency surgery.
* Patients with severe concomitant diseases and estimated survival time ≤ 5 years.
* Allergic to any component of the therapy.
* Patients with poorly differentiated adenocarcinoma, signet ring cell carcinoma, or mucinous adenocarcinoma.
* Patients who received immunosuppressive or systemic hormone therapy for immunosuppressive purposes within 1 month prior to the initiation of therapy.
* Patients who have received any other experimental drug (including immunotherapy) or participated in another interventional clinical trial within 30 days before screening.
* Factors leading to study termination, such as alcoholism, drug abuse, other serious illnesses (including psychiatric disorders) requiring combination therapy, and patients with severe laboratory abnormalities.
* Patients with congenital or acquired immune deficiency (such as HIV infection).
* Vulnerable groups, including mentally ill, cognitively impaired, critically ill patients, minors, pregnant or lactating women, illiterate, etc.

Other conditions that investigators consider not suitable for this study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Estimated)
Dates: Start 2024-02-05 (Actual); Primary Completion 2027-09-01 (Estimated); Study Completion 2028-09-01 (Estimated)

PRIMARY OUTCOMES:
Complete response | within 10 days after TNT therapy or surgery
  Pathological complete response (pCR) ：absence of residual tumour on resected specimen. Clinical complete response（cCR）: no residual tumour visible on imaging or colonoscopy and biopsy.

SECONDARY OUTCOMES:
Tumor regression grade | within 10 days after surgery
  TRG is evaluated according to the AJCC system. TRG0-1 is defined as good response, TRG2 as moderate response, and TRG3 as poor response.
Local recurrence rate(LRR) | 3 years after sugery
  Presence of adenocarcinoma within the rectal wall or within the mesorectum confirmed by pathology.
Disease free survival(DFS) | 3 years after treatment
  the time from randomization to recurrence of tumor or death
Overall survival(OS) | 3 years after enrollment
  the time from randomization to death
Adverse effects rate | From date of initiation of treatment until the date of death from any cause, assessed up to 5 years
  Rate of radiotherapy, chemotherapy and immunotherapy related adverse events
Rectal specific quality of life assessment via QLQ-CR29 | Baseline and months 3, 6, 12, 24, 36, 60 after the TNT treatment or surgery
  Rectal specific quality of life according to European Organization for Research and Treatment of Cancer ( EORTC) Quality of life questionnaire QLQ-CR29. scale from 0 to 100, A higher scale represents better function and a higher quality of life.
Quality of life assessment via QLQ-C30 | Baseline and months 3, 6, 12, 24, 36, 60 after the TNT treatment or surgery
  Quality of life according to EORTC Quality of life Questionnaire QLQ-C30 version 3.0. Score range from 0 to 100 points. A higher score represents better function and a higher quality of life.
Validation of the Wexner score | Months 3, 6, 12, 24, 36, 60 after the TNT treatment or surgery
  The change of severity of fecal incontinence assessment according to Wexner score. a score from 0-20, where 0 is perfect continence and 20 is complete incontinence.

CONTACTS AND LOCATIONS:
Locations (1):
- Zhejiang University Affiliated Jinhua Hospital, Jinhua, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Yes
JinhuaCH will share de-identified individual data that underlie the results reported. A decision concerning the sharing of other study documents, including protocol and statistical analysis plan will be examined upon request.
Supporting Information: Study Protocol, SAP
Time Frame: inhuaCH will consider access to study data upon a written detailed request sent to JinhuaCH, from 6 months until 5 years after publication of summary data.
Access Criteria: The data shared will be limited to that required for independent mandated verification of the published results, the applicant will need authorization from JinhuaCH for personal access, and the data will only be transferred after signing of a data access agreement.
URL: http://www.jhzxyy.cn/